CLINICAL TRIAL: NCT04679519
Title: The Effects of Protein Supplementation in Females and Males Following Acute Eccentric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/SPS/007
Record Dates: First submitted 2020-12-10; First posted 2020-12-22 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Muscle Damage

STUDY DESIGN:
Intervention Model Description: Randomised control study with four groups, one control and three protein supplements.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Control group that was not given a supplement.
  Interventions: Other: Drop Jumps
- BCAA (Experimental): Supplement group that was given Branched Chain Amino Acids (BCAA).
  Interventions: Other: Drop Jumps
- Leucine (Experimental): Supplement group that was given Leucine.
  Interventions: Other: Drop Jumps
- HMB (Experimental): Supplement group that was given β-Hydroxy β-methylbutyric acid (HMB)
  Interventions: Other: Drop Jumps

INTERVENTIONS:
Other: Drop Jumps — Perform 100 drop jumps from 40 cm height. The protocol is divided into 5 sets of 20 repetitions. Between each repetition participants get 10 seconds, and between each set 2 minutes rest. Stand on the box, drop of the box and land with feet shoulder width apart. Then immediately bend knee to approx 45 degrees and jump straight up. Throughout each jump hands are placed on hips and should not move.

SUMMARY:
Examine the impact of the protein supplements leucine, HMB and BCAA on muscle recovery and inflammatory response following acute exercise.

DETAILED DESCRIPTION:
Participants, both females and males, will perform an acute bout of exercise. A bout of exercise that will involve multiple drop jumps. Prior to and post exercise, functional outputs will be measured and blood will be collected to quantify the inflammatory response. The protocol will involve attending the laboratory on 6 occasions over a two week period to complete the above measures.

ELIGIBILITY:
Inclusion Criteria:

* Health recreationally active males and females.

Exclusion Criteria:

* Asthma sufferers
* People with kidney disease
* People partaking in lower limb strength training
* People suffering DOMS in the past 6 months
* People already taking dietary supplements, other NSAIDs, or for example aspirin, alcohol, warfarin, phenytoin, methotrexate, lithium, diuretics, cyclosporine.
* People with bone or soft tissue injury within last 12 months
* People with gastric problems
* People with hypertension
* People who have had history of heart failure
* People with liver disease
* People with connective tissue disorders
* People with Crohn's disease
* People with ulcerative colitis
* People with peripheral arterial disease
* People with cerebrovascular disease
* Elderly population
* People with allergies to NSAIDs, Omega- 3 fatty acids and BCAAs.
* People with depression
* People with bipolar disorder
* People with diabetes
* Females who are pregnant
* People who have HIV / AIDS

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Concentration of Creatine Kinase at baseline | Baseline
  Blood taken from either vein or finger will be analysed for creatine kinase, a marker of muscle damage.
Concentration of Creatine Kinase immediately after intervention. | Immediately after intervention.
  Blood taken from either vein or finger will be analysed for creatine kinase, a marker of muscle damage.
Concentration of Creatine Kinase at 24 hours after intervention. | 24 hours after intervention.
  Blood taken from either vein or finger will be analysed for creatine kinase, a marker of muscle damage.
Concentration of Creatine Kinase at 48 hours after intervention. | 48 hours after intervention.
  Blood taken from either vein or finger will be analysed for creatine kinase, a marker of muscle damage.
Concentration of Creatine Kinase at 7 days after intervention. | 7 days after intervention.
  Blood taken from either vein or finger will be analysed for creatine kinase, a marker of muscle damage.
Concentration of Creatine Kinase at 14 days after intervention. | 14 days after intervention.
  Blood taken from either vein or finger will be analysed for creatine kinase, a marker of muscle damage.
Number of Chair Rises at baseline | Baseline
  Stand and sit on chair consecutively for 30 seconds with hands placed on hips.
Number of Chair Rises immediately after intervention. | Immediately after intervention.
  Stand and sit on chair consecutively for 30 seconds with hands placed on hips.
Number of Chair Rises at 24 hours after intervention. | 24 hours after intervention.
  Stand and sit on chair consecutively for 30 seconds with hands placed on hips.
Number of Chair Rises at 48 hours after intervention. | 48 hours after intervention.
  Stand and sit on chair consecutively for 30 seconds with hands placed on hips.
Number of Chair Rises at 7 days after intervention. | 7 days after intervention.
  Stand and sit on chair consecutively for 30 seconds with hands placed on hips.
Number of Chair Rises at 14 days after intervention. | 14 days after intervention.
  Stand and sit on chair consecutively for 30 seconds with hands placed on hips.
Squat Jump height at baseline | Baseline
  Hands placed on hips, feet shoulder width apart. Bend knees to approx 45 degrees hold for 3 seconds and jump maximally.
Squat Jump height immediately after intervention. | Immediately after intervention.
  Hands placed on hips, feet shoulder width apart. Bend knees to approx 45 degrees hold for 3 seconds and jump maximally.
Squat Jump height at 24 hours after intervention. | 24 hours after intervention.
  Hands placed on hips, feet shoulder width apart. Bend knees to approx 45 degrees hold for 3 seconds and jump maximally.
Squat Jump height at 48 hours after intervention. | 48 hours after intervention.
  Hands placed on hips, feet shoulder width apart. Bend knees to approx 45 degrees hold for 3 seconds and jump maximally.
Squat Jump height at 7 days after intervention. | 7 days after intervention.
  Hands placed on hips, feet shoulder width apart. Bend knees to approx 45 degrees hold for 3 seconds and jump maximally.
Squat Jump height at 14 days after intervention. | 14 days after intervention.
  Hands placed on hips, feet shoulder width apart. Bend knees to approx 45 degrees hold for 3 seconds and jump maximally.
Range of motion at baseline. | Baseline
  Sit on chair, then flex and extend legs three times from 90 degrees position.
Range of motion immediately after intervention. | Immediately after intervention.
  Sit on chair, then flex and extend legs three times from 90 degrees position.
Range of motion at 24 hours after intervention. | 24 hours after intervention.
  Sit on chair, then flex and extend legs three times from 90 degrees position.
Range of motion at 48 hours after intervention. | 48 hours after intervention.
  Sit on chair, then flex and extend legs three times from 90 degrees position.
Range of motion at 7 days after intervention. | 7 days after intervention.
  Sit on chair, then flex and extend legs three times from 90 degrees position.
Range of motion at 14 days after intervention. | 14 days after intervention.
  Sit on chair, then flex and extend legs three times from 90 degrees position.
Inflammatory cytokines concentration at baseline | Baseline
  Blood from vein will be analysed for 10 different cytokines. Different cytokines include interleukins 1 beta, 2, 3, 4, 7, 8, 10, 17 and tutor necrosis factor receptor 1.
Inflammatory cytokines concentration at 24 hours after intervention. | 24 hours after intervention.
  Blood from vein will be analysed for 10 different cytokines. Different cytokines include interleukins 1 beta, 2, 3, 4, 7, 8, 10, 17 and tutor necrosis factor receptor 1.
Inflammatory cytokines concentration at 48 hours after intervention. | 48 hours after intervention.
  Blood from vein will be analysed for 10 different cytokines. Different cytokines include interleukins 1 beta, 2, 3, 4, 7, 8, 10, 17 and tutor necrosis factor receptor 1.
Inflammatory cytokines concentration at 7 days after intervention. | 7 days after intervention.
  Blood from vein will be analysed for 10 different cytokines. Different cytokines include interleukins 1 beta, 2, 3, 4, 7, 8, 10, 17 and tutor necrosis factor receptor 1.
Concentration of Lactate from baseline to immediately after intervention. | Baseline and immediately after intervention.
  Blood drop from finger will be used to lactate.
Muscle Soreness | Daily for 14 days.
  Record soreness on visual analogue scale from 1-10 1 = low soreness, 10 = extreme soreness.

SECONDARY OUTCOMES:
Weighed food diaries. | Daily for 14 days.
  Fill out dietary intake on food diary, by weighing food.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participant data to be published.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Howatson G, Hoad M, Goodall S, Tallent J, Bell PG, French DN. Exercise-induced muscle damage is reduced in resistance-trained males by branched chain amino acids: a randomized, double-blind, placebo controlled study. J Int Soc Sports Nutr. 2012 Jul 12;9:20. doi: 10.1186/1550-2783-9-20. eCollection 2012. PMID 22569039
- [Background] Kirby TJ, Triplett NT, Haines TL, Skinner JW, Fairbrother KR, McBride JM. Effect of leucine supplementation on indices of muscle damage following drop jumps and resistance exercise. Amino Acids. 2012 May;42(5):1987-96. doi: 10.1007/s00726-011-0928-9. Epub 2011 May 12. PMID 21562819